CLINICAL TRIAL: NCT01698931
Title: Efficacy of Repaglinide Compared to Glyburide and Placebo on Hepatic Glucose Metabolism in Type 2 Diabetic Subjects Treated With Diet or With Antidiabetic Oral Agents. A Randomized, Open, Cross-over Single-centre Placebo-controlled Trial
Brief Title: Efficacy of Repaglinide in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AGEE-1259
Record Dates: First submitted 2012-10-01; First posted 2012-10-03 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — repaglinide; Glyburide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment period 1 (Experimental)
  Interventions: Drug: repaglinide; Drug: glyburide; Drug: placebo
- Treatment period 2 (Active Comparator)
  Interventions: Drug: repaglinide; Drug: glyburide; Drug: placebo
- Treatment period 3 (Placebo Comparator)
  Interventions: Drug: repaglinide; Drug: glyburide; Drug: placebo

INTERVENTIONS:
Drug: repaglinide — 1 mg before each main meal on three separate dosing visits separated by a wash-out period
Drug: glyburide — 5 mg before breakfast and before supper on three separate dosing visits separated by a wash-out period
Drug: placebo — Before each main meal on three separate dosing visits separated by a wash-out period

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to compare the efficacy of repaglinide to glyburide and placebo on hepatic glucose metabolism in subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* HbA1c (glycosylated haemoglobin A1c) above 7 %
* BMI (body mass index) below 32 kg/m^2
* FBG (fasting blood glucose) after wash out period 130-220 mg/dl
* Currently treated with diet or OHA (oral hypoglycaemic agent)

Exclusion Criteria:

* Current systemic treatment with concomitant medication
* Known or suspected history of drug or alcohol dependence
* Any other significant concomitant disease such as cerebrovascular or symptomatic peripheral vascular disease, malignant, disease or severe treated or untreated hypertension
* Hepatic disease
* Cardiac problems
* Active proliferative retinopathy
* Known or suspected allergy to trial product or related products
* Women in fertile age and women having the intention of becoming pregnant
* Body Mass Index (BMI) above 32 kg/m^2

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2002-04-26 (Actual); Primary Completion 2003-03-06 (Actual); Study Completion 2003-03-06 (Actual)

PRIMARY OUTCOMES:
Basal hepatic glucose production | Day 0; day 44

SECONDARY OUTCOMES:
Number of hypoglycaemic episodes | Day 0; day 44
Change in body weight | Day 0; day 44
Number of adverse events | Day 0; day 44

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Padua, Italy

REFERENCES:
- [Result] Ciccarone A, Mari A, Pulizzi N, Bianchi C, Palumbo F, Benzi L, Del Prato S. Assessment of insulin secretion in response to a mixed meal in type 2 diabetes. Effects of short-term repaglinide and glibenclamide administration. Diabetologia 2005; 48 (Suppl. 1): A284 (Abstract No. PS65-781)
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com